CLINICAL TRIAL: NCT00000931
Title: A Randomized Clinical Trial of the Efficacy of a Behavioral Intervention to Prevent Acquisition of HIV Among Men Who Have Sex With Men
Brief Title: HIV Prevention Counseling for Men Who Have Sex With Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Prevention
Other Study IDs: HIVNET 015
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2006-11

CONDITIONS: HIV Infections
Keywords: Homosexuality, Male; Risk-Taking; Behavior Therapy; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality, Male; Risk-Taking | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavioral intervention
Behavioral: Risk-reduction counseling

SUMMARY:
The purpose of this study is to see if a behavioral intervention, a special kind of counseling, can reduce the risk of HIV infection in men who have sex with men. The behavioral intervention will be compared to the standard risk reduction counseling that is given before and after getting an HIV test.

In standard pre- and post-test counseling, everyone is told the same things about how to prevent HIV. The behavioral intervention used in this study is designed to help each individual prevent HIV according to his specific problems and needs.

DETAILED DESCRIPTION:
The intervention being evaluated in this trial is based on the extensive literature on behavioral approaches to risk reduction in MSM. These reviews recommend an intervention that, unlike the current standard HIV pre-test and post-test risk-reduction counseling, is tailored to an individual's unique problems and needs, lifestyle, and situations that contribute to high-risk behavior. Furthermore, there is a need for HIV-prevention intervention trials using biological endpoints (e.g., HIV seroconversion) in addition to behavioral change indices.

Participants are randomly assigned to receive either the behavioral intervention or the control risk-reduction counseling. The same counseling staff provides the two types of treatment. The behavioral intervention consists of 10 counseling sessions within a 4-month period followed by quarterly maintenance sessions for the remainder of the 3-year follow-up. The intervention is conducted on a one-to-one basis and targets condom use, change in sexual practices associated with HIV risk, and change in sexual practices in the context of alcohol and drug use. Participants in the control group receive pre- and post-test counseling at enrollment, then semiannually through Month 36. Beginning at Month 6, all participants complete routine semiannual visits. At each visit, Risk Assessment and phlebotomy for specimen collection for HIV antibody tests are administered. As is routine in most public counseling and testing venues, participants in the control condition do not see the same counselor consistently.

ELIGIBILITY:
Inclusion Criteria

Participants may be eligible for this study if they:

* Are an HIV-negative man who has had anal sex with another man in the 12 months prior to study entry.
* Are able to attend all scheduled study visits.
* Are able to provide information for locator purposes (address, phone number, etc.).
* Are at least 18 years old.

Exclusion Criteria

Participants will not be eligible for this study if they:

* Have been in a monogamous relationship for 2 years or more with an HIV-negative man. (Monogamous is defined as a relationship in which the members of the couple engage in sexual activities with only each other.)
* Have an obvious mental disorder or any another condition that would prevent them from completing the study.
* Are currently enrolled in any Phase III HIV vaccine trial, including the AIDSVAX Phase III trial sponsored by VaxGen, Inc.
* Are currently enrolled in HIVNET Protocol 014.
* Were enrolled in the HIVNET 015 Pilot Study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4350

CONTACTS AND LOCATIONS:
Overall Officials: Chesney M, Coates T, Study Chair; Koblin B, Study Chair
Locations (6):
- United States (6):
  - San Francisco Dept of Hlth / AIDS Office, San Francisco, California
  - Denver Dept of Public Health / HIVNET, Denver, Colorado
  - Howard Brown Health Ctr, Chicago, Illinois
  - Fenway Community Health Ctr, Boston, Massachusetts
  - New York Blood Ctr, The Bronx, New York
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Result] Koblin B, Chesney M, Coates T; EXPLORE Study Team. Effects of a behavioural intervention to reduce acquisition of HIV infection among men who have sex with men: the EXPLORE randomised controlled study. Lancet. 2004 Jul 3-9;364(9428):41-50. doi: 10.1016/S0140-6736(04)16588-4. PMID 15234855